CLINICAL TRIAL: NCT00809432
Title: Beneficial Cardiovascular Effects of Reducing Exposure to Particulate Air Pollution With a Simple Facemask
Brief Title: The Cardiovascular Benefits of Reducing Personal Exposure to Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Professor David E Newby, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 167/2008/Pilot
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Blood Pressure; Heart Rate Variability
Keywords: Air pollution; Heart rate; Heart rate variability; Blood pressure; Face mask
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visit 1 (Experimental): 2 hour city centre kerbside walk in Beijing China
  Interventions: Other: No Face mask
- Visit 2 (Experimental): 2 hour city centre kerbside walk in Beijing China
  Interventions: Device: Face mask (Dust Respirator)

INTERVENTIONS:
Device: Face mask (Dust Respirator) — Subjects to wear a simple face mask for 24 hours prior to the study day and the 24 hours of the study day. They will be instructed to wear the mask as much as possible when indoors and at all times when outdoors.
  Other Names: 3M Dust Respirator 8812
  Arms: Visit 2
Other: No Face mask — Subjects will not wear a face mask to reduce their personal exposure to air pollution
  Arms: Visit 1

SUMMARY:
Exposure to air pollution is an important risk factor for cardiovascular morbidity and mortality, and is associated with increased blood pressure, reduced heart rate variability, endothelial dysfunction and myocardial ischaemia. The study objectives were to assess the potential cardiovascular benefits of reducing personal particulate air pollution exposure by wearing a facemask in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Current smokers
* Significant occupational exposure to air pollution
* Regular medication use (except oral contraceptive pill)
* Intercurrent illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | During 24 hour study period

SECONDARY OUTCOMES:
Heart rate | During 24 hour study period
Heart rate variability | During 24 hour study period
Personal air pollution exposure | During 2 hour city centre walk

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Langrish, MB BCh MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Medical Union College, Beijing, China

REFERENCES:
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535